CLINICAL TRIAL: NCT05947123
Title: Real-life Study of the Efficacy of Management of Migraine Patients After Failure of 2 Prophylactic Treatments: a Retrospective Study
Brief Title: Real-life Study of the Efficacy of Management of Migraine Patients After Failure of 2 Prophylactic Treatments
Acronym: EVIREMIG
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-07Obs-CHRMT
Record Dates: First submitted 2023-07-07; First posted 2023-07-17 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Migraine
Keywords: migraine; prophylactic treatment; real life
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Patient health care observational follow up after 2 prophylactic tratments — Real-life, observational, single-center cohort study to describe the efficacy of prophylactic treatment in patients after failure of at least 2 prophylactic treatments. Patients included in the study will be followed up in consultations or day hospitals according to their usual care, and will be asked to complete the MIDAS, HIT-6, PGIC, HAD and WPAI questionnaires at each visit. Data describing their care will be extracted from computerized patient records.

SUMMARY:
This is a real-life, observational, single-center cohort study to describe the efficacy of prophylactic treatment in patients after failure of at least 2 prophylactic treatments. Patients included in the study will be followed up in consultations or day hospitals according to their usual care, and will be asked to complete the MIgraine Disability Assessment (MIDAS), Headache Impact Test short-form (HIT-6), Patient Global Impression of Change (PGIC), Hospital Anxiety and Depression (HAD) scale and Work and Personal Activities Impairment (WPAI) questionnaires at each visit.

Data describing their care will be extracted from computerized patient records.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Migraine [International Headache Society (IHS) criteria 2013, revised 2018] with or without aura
* Monthly number of attacks ≥ 8 for at least 3 months
* Indication for prophylactic treatment
* For eptinezumab: resistance to at least 2 conventional disease-modifying therapies
* Agrees to use data for research purposes

Exclusion Criteria:

* Vascular history: myocardial infarction (MI), unstable angina or coronary bypass surgery, stroke or transient ischemic attack (TIA), Peripheral Arterial Disease of the Lower Limbs (PAD), uncontrolled hypertension

  * Need for analgesics for a cause other than migraine
  * Difficulty in understanding French language or cognitive impairment that compromises completion of self-questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Migraine [International Headache Society (IHS) criteria 2013, revised 2018] with or without aura
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Headache Impact Test in patients with migraine at 12 months | 12 months after prophylactic treatments
  Using HIT-6 (Headache Impact Test short-form) questionnaire which addresses six main domains affected by headaches, including pain, social functioning, role functioning, cognitive functioning, vitality and psychological stress. This survey is extremely useful for screening and monitoring how headaches affect patients in their day-to-day lives over time.
  Each item is answered on a 5-point Likert scale (6 = never, 8 = rarely, 10 = sometimes, 11 = very often, 13 = always). The scoring of the HIT-6 was derived to approximate the total score obtained from a larger battery of items, using results from item response theory (IRT) [10]. The final score is obtained from simple summation of the six items.

SECONDARY OUTCOMES:
Headache-related disability in patients with migraine at 12 months | 12 months after prophylactic treatments
  MIDAS scale (Migraine Disability Assessment) measures headache-related disability and improve doctor-patient communication about the functional consequences of migraine. The questionnaire was based on five disability questions that focus on lost time in three domains: schoolwork or work for pay; household work or chores; and family, social, and leisure activities.
  This instrument is scored as follows: 5 to 10 indicates little or no disability, 10 to 20 indicates moderate disability, and higher than 20 denotes severe disability.
Anxiety and Depression state evaluation in patients with migraine at 12 months | 12 months after prophylactic treatments
  Using Hospital Anxiety and Depression Scale (HADS) : is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score.
  The depression items tend to focus on the anhedonic symptoms of depression. Items are rated on a 4-point severity scale.
  The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states. Scores of greater than or equal to 11 on either scale indicate a definitive case.
Migraine occurence in patients with migraine at 12 months | 12 months after prophylactic treatments
  Number of migraine days
Crisis treatments in patients with migraine at 12 months | 12 months after prophylactic treatments
  Number of crisis treatments taken
Patient Global Impression of Change in patients with migraine at 12 months | 12 months after prophylactic treatments
  Using Patient Global Impression of Change (PGIC) score: a 7 point scale depicting a patient's rating of overall improvement.
  Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Work and Personal Activities Impairment in patients with migraine at 12 months | 12 months after prophylactic treatments
  Using Work and Personal Activities Impairment (WPAI) score : a well validated instrument to measure impairments in work and activities.
  WPAI scores are based on 1-item (presenteeism, activitity impairment), 2-items (absenteeism) and multiple items (overall work productivity).
Most Bothersome Symptom in patients with migraine at 12 months | 12 months after prophylactic treatments
  Most Bothersome Symptom (MBS)
Days off work at 12 months | 12 months after prophylactic treatments
  Number of days off work
Emergency room visits at 12 months | 12 months after prophylactic treatments
  Number of emergency room visits
Type of prophylactic treatment used at 12 months | 12 months after prophylactic treatments
  Type of prophylactic treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DUCROCQ, MD, Principal Investigator — CHR Metz Thionville Hopital de Mercy
Locations (1):
- CHR Metz-Thionville/Hopital de Mercy, Metz, France

IPD SHARING:
Plan to Share IPD: No